CLINICAL TRIAL: NCT06791837
Title: Cerebral Lactate Uptake and Transport in Obese and Non-Obese Individuals
Brief Title: Brain Blood Flow and Lactate in Non-obese and Obese Subjects
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Other Study IDs: 2125746
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabetes; Obesity
Keywords: lactate; obesity; exercise
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-obese: individuals with a BMI<25 kg/m2
  Interventions: Behavioral: EXERCISE
- obese: individuals with a BMI 30-40 kg/m2
  Interventions: Behavioral: EXERCISE

INTERVENTIONS:
Behavioral: EXERCISE — each group will undergo a max test and a submaximal exercise test

SUMMARY:
Cerebral blood flow (CBF) is essential for maintaining brain health and function, as it ensures delivery oxygen and nutrients necessary to support neuronal activity. Reduced CBF can impair the brain's ability to meet its metabolic demands, leading to deficits in cognitive ability. Impairments in CBF are associated with cognitive decline and neurodegenerative disease such as Alzheimer's and dementia. Many factors influence CBF, but recently lactate has emerged as a key player. Blood glucose has long been considered the primary fuel for the brain, but emerging evidence indicates that lactate may be the preferred fuel for neurons, and lactate may become even more important under stressful conditions.

Individuals with obesity often have impaired lactate metabolism resulting in higher resting blood lactate concentrations and reduced ability to clear lactate after a physiological stress. At the same time, it is known that exercise is a powerful intervention for improving lactate metabolism.

Thus, this project seeks to investigate the role of lactate in brain blood flow in individuals with and without obesity as well as establish if short term exercise training (individuals with obesity only) will alter circulating lactate concentrations at rest and in response to exercise.

DETAILED DESCRIPTION:
Blood lactate is often considered a waste product from aerobic metabolism. Many people assume it causes fatigue and muscle. Lactate is a signaling molecule in the body. In addition lactate is also a fuel. Evidence supports that lactate may be more important when the brain is stressed. We also know that individuals with obesity and/or type 2 diabetes may have impaired lactate metabolism.

The investigators will compare brain blood flow and lactate response to an exercise stress test and submaximal exercise in obese and non-obese individuals.

ELIGIBILITY:
Inclusion Criteria:

healthy adult men and women 18-45 years of age BMI 18-40 kg/m2 not pregnant, premenopausal with regular menstrual cycles not breastfeeding non-nicotine users

Exclusion Criteria:

medications known to affect sleep, autonomic control, blood lactate levels or metabolic, or cardiovascular function (PI discretion) self-reported history of hepatic, renal, pulmonary, cardiovascular, or neurological disease, stroke or neurovascular disease, bleeding/clotting disorders, sleep apnea or other sleep disorders, diabetes, history of alcoholism or substance abuse major cardiovascular event or surgical procedure within the past three months hypertension (>140/90 mmHg or at PIs discretion).

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals that live in the area of Columbia, MO
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
brain blood flow | over the 30 minutes of testing
  Using transcranial doppler we will measure brain blood flow

SECONDARY OUTCOMES:
lactate concentrations | over ~ 60 minutes of testing
  Lactate will be measured in response to an exercise stress test as well as to a submaximal exercise bout

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
only coded IPD will be shared that is used in the results published
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication and ending 5 yr after publication of results
Access Criteria: Mean data will be shared for meta analysis For access to individual data, a proposal that described the planned analysis must be submitted and an agree must be signed by the applicant. These documents would be submitted to the PI.
URL: https://clinicaltrials.gov/policy/protocol-definitions?popup=true#IPDSharingAccess

REFERENCES:
- [Background] Xue X, Liu B, Hu J, Bian X, Lou S. The potential mechanisms of lactate in mediating exercise-enhanced cognitive function: a dual role as an energy supply substrate and a signaling molecule. Nutr Metab (Lond). 2022 Jul 30;19(1):52. doi: 10.1186/s12986-022-00687-z. PMID 35907984
- [Background] Bouzier-Sore AK, Voisin P, Canioni P, Magistretti PJ, Pellerin L. Lactate is a preferential oxidative energy substrate over glucose for neurons in culture. J Cereb Blood Flow Metab. 2003 Nov;23(11):1298-306. doi: 10.1097/01.WCB.0000091761.61714.25. PMID 14600437
- [Background] Brooks GA, Osmond AD, Arevalo JA, Duong JJ, Curl CC, Moreno-Santillan DD, Leija RG. Lactate as a myokine and exerkine: drivers and signals of physiology and metabolism. J Appl Physiol (1985). 2023 Mar 1;134(3):529-548. doi: 10.1152/japplphysiol.00497.2022. Epub 2023 Jan 12. PMID 36633863
- See also: background information — https://pmc.ncbi.nlm.nih.gov/articles/PMC5315230/